CLINICAL TRIAL: NCT06835101
Title: The Effect of Music Versus Midazolam on Perioperative Anxiety of Obese Patients Under Spinal Anesthesia
Brief Title: Perioperative Music in Obese Patients Under Spinal Anesthesia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asklepieion Voulas General Hospital (Other Government)
Responsible Party: Principal Investigator, Maria Diakomi, Consultant Anaesthesiologist, General Hospital of Kavala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 25870/9-10-24
Record Dates: First submitted 2025-01-15; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Obesity, Adolescent
Keywords: obese; music; anxiety
MeSH Terms: conditions — Pediatric Obesity; Obesity; Anxiety Disorders | interventions — Midazolam; Hypnotics and Sedatives

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Music group (Active Comparator): The "music" group will receive music beginning 20 minutes before spinal anesthesia until the end of surgery.
  Interventions: Other: Music intervention
- Midazolam group (Active Comparator): The "midazolam" group will receive increments of midazolam beginning 20 minutes before spinal anesthesia.
  Interventions: Drug: Midazolam (sedative)

INTERVENTIONS:
Other: Music intervention — The "music" group will receive music beginning 20 minutes before spinal anesthesia until the end of surgery.
  Arms: Music group
Drug: Midazolam (sedative) — The "midazolam" group will receive increments of midazolam beginning 20 minutes before spinal anesthesia.
  Arms: Midazolam group

SUMMARY:
The goal of this clinical trial is to learn whether music or midazolam has a greater anxiolytic effect on obese patients undergoing spinal anesthesia. It will also determine the safety of music compared to midazolam in this population (differences in blood pressure, heart rate, oxygen saturation). The main question to answer: Music or midazolam is more effective in reducing anxiety in obese patients under spinal anesthesia?

ELIGIBILITY:
Inclusion Criteria:

* patients who are > 18 years old
* patients with Body Mass Index -ΒΜΙ>30 kg/m2
* patients who will give informed consent in receiving spinal anaesthesia
* patients who will give informed consent in participating in the study

Exclusion Criteria:

* absolute contraindications of spinal anaesthesia,
* severe psychiatric, cognitive or sensory impairment
* mother language other than greek,
* known hypersensitivity to midazolam,
* renal impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Spielberger State-Trait Anxiety Inventory (STAI): State -anxiety immediately after spinal anesthesia. | State -anxiety is measured immediately after spinal anesthesia.
  State -anxiety, how the person feels at the moment, is measured by means of Spielberger State-Trait Anxiety Inventory (STAI).
  STAI tool scores range from 20 to 80, with higher scores indicating higher anxiety. Although it is difficult to represent severity of anxiety with a numerical cut-off, a score of 50 or higher has been shown to be associated with a higher level of anxiety.

SECONDARY OUTCOMES:
Spielberger State-Trait Anxiety Inventory (STAI): State -anxiety immediately after surgery | Immediately after surgery
  State -anxiety, how the person feels at the moment, is measured by means of Spielberger State-Trait Anxiety Inventory (STAI).
  STAI tool scores range from 20 to 80, with higher scores indicating higher anxiety. Although it is difficult to represent severity of anxiety with a numerical cut-off, a score of 50 or higher has been shown to be associated with a higher level of anxiety.
Time performing spinal anesthesia | From the start of positioning maneuvers for spinal anesthesia to the spinal needle removal
  Time needed for spinal anesthesia performance, measured in minutes
Patient satisfaction 24 hours after surgery | 24 hours after surgery
  The patient will be asked 24 hours after surgery whether he/she is satisfied (yes/no) with anesthesia.
Communication difficulties between the patient and the anesthesiologist. | Immediately after surgery
  The patient will be asked if there was any problem communicating with the anesthesiologist.
Communication difficulties between the anesthesiologist and the patient. | Immediately after surgery
  The anesthesiologist will record any difficulty in communication with the patient during spinal anesthesia.
Adverse outcomes | During the operation
  Any adverse outcome during the operation will be recorded.

CONTACTS AND LOCATIONS:
Locations (3):
- Greece (3):
  - Asklepieion Hospital of Voula, Athens, Voula
  - General Hospital of Kavala, Kavala
  - General Hopsital of Rethymno, Rethymno